CLINICAL TRIAL: NCT01486160
Title: Etiology, Frequency and Epidemiology of Respiratory Viral Infection in Nursing Home Residents
Brief Title: Respiratory Viral Infection in Nursing Home Slovenia
Status: Completed | Type: Observational
Sponsor: University Maribor (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other); University Medical Centre Maribor (Other); University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Nina Gorisek Miksic, Nina Gorisek Miksic, MD, M.Sc, infectologist, University Maribor
Other Study IDs: DSO-2011-2012
Record Dates: First submitted 2011-12-01; First posted 2011-12-06 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Acute Viral Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- nursing home residents: participants in this group are nursing home residents
- Nursing home employees: Participants in this group are health care workers, employees at the nursing home

SUMMARY:
This study will be conducted in a 208-bed nursing home in Maribor. The investigators will observe a group of a 100 nursing-home residents and 50 health care workers- employees in the nursing home- in a six months period.Influenza vaccination status will be recorded in all participants at the beginning.

At the beginning and at the end of the study the blood samples for vitamin D concentration determination and nasopharyngeal swabs for molecular detection of respiratory viruses will taken in all of the participants.

The study will observe number of viral respiratory tract infection in participants and identify the viral etiology of infections during 6 months observational period.Nasopharyngeal swab and blood sample will be taken in each of the participant who will suffer an acute respiratory tract infection (upper or lower respiratory tract infection) and viral agents of respiratory tract diseases will be searched for. The investigators will try to detect different viral agents of respiratory tract infection: human rhinoviruses, enteroviruses, influenza A, B, parainfluenza 1-4, respiratory syncytial virus, human coronaviruses, human metapneumovirus, adenoviruses and human bocavirus with newer molecular methods (real-time polymerase chain reaction, real-time reverse transcriptase polymerase chain reaction) in nasopharyngeal swab and in blood sample of the participants.

During the study period the investigators will monitor the daily number of visitors (adults, preschool children and pupils) in each nursing home room. The epidemiological aspect of respiratory viral infection will be assessed.

Our study hypothesis is that lower respiratory tract infections in elderly can be caused by viruses other than influenza.

The investigators would like to know if hypovitaminosis D is a risk factor for respiratory tract infections in nursing home residents and employees.

The investigators would also like to know if the number of respiratory tract infections in elderly correlates with the number of visitors in nursing home, small children in particular.

ELIGIBILITY:
Inclusion Criteria:

* resident of the nursing home or employee ni the nursing home

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing home residents and employees of the nursing home
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of viral respiratory tract infection in participants according to etiology | 6 months
  Number of participants with upper and lower respiratory tract infection will be detected and etiology of viral infection will be identified

SECONDARY OUTCOMES:
Serum vitamine D concentration in participants | 6 months
  Serum concentration of vitamine D will be measured retrospectively from the blood samples taken at the beginning of the study and correlation between vitamine D concentration and the frequency of respiratory tract infection in participants will be made
Daily number of visitors in nursing home in correlation with the number of respiratory tract infection in residents | 6 months
  Daily number of visitors in each nursing home room will be counted and correlate with the number of respiratory tract infection in participants.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Gorisek Miksic, MD, M.sc, Principal Investigator — University Medical Centre Maribor
Locations (1):
- Nursing home Tezno, Maribor, Maribor City Municipality, Slovenia

REFERENCES:
- [Background] Beck-Sague C, Banerjee S, Jarvis WR. Infectious diseases and mortality among US nursing home residents. Am J Public Health. 1993 Dec;83(12):1739-42. doi: 10.2105/ajph.83.12.1739. PMID 8259806
- [Result] Mahony JB. Detection of respiratory viruses by molecular methods. Clin Microbiol Rev. 2008 Oct;21(4):716-47. doi: 10.1128/CMR.00037-07. PMID 18854489
- [Result] Pavia AT. Viral infections of the lower respiratory tract: old viruses, new viruses, and the role of diagnosis. Clin Infect Dis. 2011 May;52 Suppl 4(Suppl 4):S284-9. doi: 10.1093/cid/cir043. PMID 21460286
- [Result] Jartti L, Langen H, Soderlund-Venermo M, Vuorinen T, Ruuskanen O, Jartti T. New respiratory viruses and the elderly. Open Respir Med J. 2011;5:61-9. doi: 10.2174/1874306401105010061. Epub 2011 Jul 6. PMID 21760867
- [Result] Laaksi I, Ruohola JP, Mattila V, Auvinen A, Ylikomi T, Pihlajamaki H. Vitamin D supplementation for the prevention of acute respiratory tract infection: a randomized, double-blinded trial among young Finnish men. J Infect Dis. 2010 Sep 1;202(5):809-14. doi: 10.1086/654881. No abstract available. PMID 20632889
- [Result] Ginde AA, Mansbach JM, Camargo CA Jr. Association between serum 25-hydroxyvitamin D level and upper respiratory tract infection in the Third National Health and Nutrition Examination Survey. Arch Intern Med. 2009 Feb 23;169(4):384-90. doi: 10.1001/archinternmed.2008.560. PMID 19237723
- [Derived] Ursic T, Miksic NG, Lusa L, Strle F, Petrovec M. Viral respiratory infections in a nursing home: a six-month prospective study. BMC Infect Dis. 2016 Nov 4;16(1):637. doi: 10.1186/s12879-016-1962-8. PMID 27814689